CLINICAL TRIAL: NCT00432289
Title: Acupuncture for Treatment of Acute Spinal Cord Injury
Brief Title: Acupuncture for Treatment of Acute Spinal Cord Injury: an Exploratory/Developmental Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Amit Jha, MD, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT002763 (NIH)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Spinal Cord Injury
Keywords: neurological function
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acupuncture — Acupunture treatment 3x per week for 6 weeks.

SUMMARY:
Specific Aim: to implement and evaluate a research protocol for demonstrating the efficacy of Acupuncture Therapy to improve neurological recovery after incomplete SCI compared to a control protocol.

Hypothesis: acupuncture treatment results in greater neurological recovery than a control treatment after an incomplete SCI.

Before conducting a larger, more definitive study, this exploratory and developmental work is focused on assessing whether blinding is possible, reproducibility of the outcome measure, determine enrollment rates and effect sizes and identify clinical resources needed to conduct a larger study.

DETAILED DESCRIPTION:
The research design for this exploratory/developmental R21 application will be the same as the anticipated design for a future definitive R01 investigation. A randomized controlled treatment study will be used to compare neurological recovery after spinal cord injury (SCI) in individuals receiving an acupuncture protocol designed to maximize treatment effectiveness (treatment protocol) with an alternative acupuncture protocol designed to minimize treatment effectiveness (control). The two acupuncture protocols will be identical except for 1) needle placement, 2) use of sham, non-penetrating needles and 3) use of electricity for needle stimulation. The two protocols are designed to be indistinguishable to an individual, so participants will remain blind to whether they are receiving the treatment or the control protocol.

Specific Aim: to implement and evaluate a research protocol for demonstrating the efficacy of Acupuncture Therapy to improve neurological recovery after incomplete SCI compared to a control protocol.

Hypothesis: acupuncture treatment results in greater neurological recovery than a control treatment after an incomplete SCI.

Before proposing a definitive R01 investigation to test this hypothesis, several preliminary steps are required and will be addressed in this feasibility study. Five objectives have been identified for the current R21 application as follows.

Objective 1 - Demonstrate that participants are unable to distinguish between treatment and control protocols, assuring participant blinding.

Objective 2 - Verify the inter-rater reliability of the primary outcome measures -the American Spinal Injury Association (ASIA) motor and sensory scores as defined by the ASIA Standards for Neurological Classification of SCI.1

Objective 3 - Collect pilot data for use in power analysis to determine the desired sample size in the definitive R01 investigation, including effect sizes, enrollment and dropout rates.

Objective 4 - Identify any unanticipated difficulties in implementing the treatment and control protocols and identify the clinical resources needed to conduct an R01 investigation.

Objective 5 - Prepare an application for an R01 definitive investigation including an operations manual for the protocol.

ELIGIBILITY:
Inclusion Criteria:

Individuals admitted to Craig Hospital immediately following initial acute care hospitalization with a primary diagnosis of acute SCI will be considered for study inclusion. Participants must give their informed consent, have medical clearance from their attending physician and meet the following inclusion criteria:

1. Incomplete spinal cord injury - ASIA grade B or C.
2. Age 16 years or older.
3. Must be admitted to Craig and enrolled in the study within 6 weeks of injury.
4. Patient must be able to tolerate lying on side for 30 minutes.
5. The expected length of stay will allow completion of the six-week study protocol.
6. Must agree to forego any acupuncture treatment other than the treatments prescribed in this protocol during the six week study period.

Exclusion Criteria:

1. Current involvement in any other clinical research trial
2. Concomitant treatment with anticoagulation medication (does not include those on prophylactic doses for deep venous thrombosis)
3. Any disease, concomitant injury, condition or treatment that interferes with the performance or interpretation of the neurological examinations.
4. Acupuncture sites obstructed by immobilization devices, where removal would be medically contraindicated.
5. Individuals with cardiac pacemakers.
6. Individual has a condition that, in the judgment of the investigator, precludes successful participation in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
ASIA Standards for Neurological Classification of SCI | Baseline and 6 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amit Jha, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States